CLINICAL TRIAL: NCT05675644
Title: Drospirenone for Emergency Contraception: a Dose-finding Pilot Study
Brief Title: Drospirenone-only Pill as Emergency Contraception
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22-2178
Record Dates: First submitted 2022-12-12; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2022-12

CONDITIONS: Contraception
Keywords: drospirenone; emergency contraception

STUDY DESIGN:
Intervention Model Description: 3x3 adaptive dose-finding design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose finding (Experimental): Drospirenone-only pill single-dose ranging from 16mg to 32mg
  Interventions: Drug: Drospirenone-only pill
- Primary ovulation inhibition testing (Experimental): Drospirenone-only pill single-dose at dose determined by dose finding arm
  Interventions: Drug: Drospirenone-only pill

INTERVENTIONS:
Drug: Drospirenone-only pill — Single dose based on adaptive dose-finding design

SUMMARY:
Emergency contraception (EC) provides an additional measure to help prevent pregnancy after unprotected intercourse or contraceptive failure. The two currently available oral emergency contraceptive methods, levonorgestrel (LNG) and ulipristal acetate (UPA), have differing availability and effectiveness. Overweight and obesity are strong risk factors for failure of EC containing LNG and UPA for body mass index (BMI) ≥ 26kg/m2 and ≥35kg/m2, respectively, resulting in limited EC options for much of the population. Drospirenone is a unique progestin that effectively inhibits ovulation when taken daily as progestin-only oral contraception and has pharmacokinetic properties that make it a good candidate for a novel effective emergency contraceptive method across BMI categories.

The investigators propose a dose-finding, adaptive-design pilot study evaluating if a single dose of drospirenone can inhibit ovulation prior to the luteinizing hormone (LH) surge. The dose-finding study design will be conducted in a well-established 3+3 model with 2 planned study arms stratified by BMI. The investigators hypothesize that a single dose of drospirenone will effectively inhibit ovulation when administered prior to the LH surge. This pilot data will directly support the dose selection for future research further evaluating the efficacy of drospirenone-only EC aimed at ultimately increasing oral EC options, particularly for patients with overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Overall good general health.
2. Age 18-35 years at time of enrollment.
3. BMI

   1. Initial dose-finding cohort: BMI < 30 kg/m2; thereafter no BMI limit
4. Intact uterus with at least 1 ovary.
5. Regular menstrual cycles that occur every 21-35 days:

   1. If patient is postpartum or post-second trimester abortion, she must have 3 menses (2 cycles) prior to enrollment.
   2. If patient had a first trimester abortion or pregnancy loss, she must have one spontaneous menses prior to enrollment.
6. Negative urine pregnancy test at screening visit and at time of drospirenone administration.
7. Consistent use of a barrier method or other non-hormonal birth control method throughout the study, or otherwise not at risk for pregnancy.
8. Ovulatory as confirmed by a documented screening progesterone (P4) level ≥3ng/ml at screening visit.
9. Willingness and ability to abstain from medications and supplements known to induce/inhibit CYP3A4 during the study period
10. Willingness and ability to comply with the protocol requirements.
11. Lives within the study site catchment area or within a reasonable distance from the site.

Exclusion Criteria:

1. Have a known hypersensitivity or contraindications to drospirenone.
2. Currently taking any known CYP3A4 inducers/inhibitors.
3. Medical conditions that affect liver function (e.g., hepatitis, cirrhosis; assessed via participant self-report).
4. Medical conditions that affect kidney function (e.g., chronic kidney disease, primary renal disease; assessed via participant self-report) or use of medications that can affect kidney function and/or electrolyte balance (e.g., ACE inhibitors, diuretic medications; assessed via participant self-report).
5. A known history of or presence of hyperkalemia (potassium ≥4.5mEq/L) or renal impairment (creatinine of ≥1.1mg/dL) at screening visit.
6. Known or suspected current alcohol dependence syndrome or any illicit drug use that may affect the metabolism of the drospirenone.
7. Undiagnosed abnormal uterine/genital bleeding.
8. Uncontrolled thyroid disorder.
9. Use of long-acting injectable hormonal contraceptive within the past 6 months prior to enrollment unless the patient has had at least one spontaneous menstrual cycle since the last injection.
10. Recent use of hormonal oral, patch, intravaginal, or intrauterine contraception unless that patient has had at least one spontaneous menstrual cycle since discontinuation.
11. Currently breastfeeding or are within 30 days of discontinuing breastfeeding unless the patient has already had a menses following discontinuation.
12. Planning on undergoing major surgery during study participation.
13. Planning significant weight loss during the study related to bariatric surgery, dieting, or other causes.
14. Planning pregnancy during their anticipated months of study participation

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Serum progesterone concentration | Measured daily for the seven days immediately following administration of the drospirenone-only pill dose during the Intervention cycle (each cycle is 21-35 days)
  Serum progesterone concentration measured after drug administration
Dominant ovarian follicle ultrasound measurement | Measured daily for the seven days immediately following administration of the drospirenone-only pill dose during the Intervention cycle (cycle length 21-35 days)
  Measurement of the dominant ovarian follicle in three planes (width, length, height) using transvaginal ultrasound

SECONDARY OUTCOMES:
Serum potassium concentration | Measured on the first and second days immediately following administration of the drospirenone-only pill dose during the Intervention cycle (cycle length 21-35 days)
  Measured as a safety outcome

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No